CLINICAL TRIAL: NCT06771843
Title: Kisoboka: Reducing Hazardous Alcohol Use and Optimizing Treatment as Prevention Among Men Living With HIV in Risk Environments
Brief Title: Reducing Hazardous Alcohol Use and Optimizing Treatment as Prevention Among Men Living With HIV in Risk Environments
Acronym: Kisoboka
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Makerere University Walter Reed Program (Unknown); Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: HS-2024-0086; R01AA031650 (NIH)
Record Dates: First submitted 2025-01-09; First posted 2025-01-13 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: HIV Antiretroviral Therapy (ART) Adherence; Alcohol Abuse; HIV Infection; Alcohol Use Disorder; HIV Infections
Keywords: behavioral economics; motivational interviewing
MeSH Terms: conditions — Alcoholism; HIV Infections | interventions — Economics, Behavioral; Motivational Interviewing; Mass Screening; Referral and Consultation

STUDY DESIGN:
Intervention Model Description: The study design is a 2x2 factorial randomized controlled trial (RCT); however, the investigators hypothesize an interaction between behavioral economics (BE) and motivational interviewing (MI), and therefore power the study to detect this interaction within the factorial design. With a statistically significant interaction between BE and MI the data would be analyzed as a 4-arm trial. Without a significant nor meaningful interaction the investigators would have additional power to examine effects for BE and MI vs S&R via a traditional factorial analysis. While a factorial design is often used when no interaction between interventions is expected, it is also especially useful to evaluate a hypothesized interaction.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Kisoboka (BE + MI and synergy) (Experimental)
  Interventions: Behavioral: Kisoboka
- Behavioral Economics (BE) (Experimental)
  Interventions: Behavioral: Behavioral Economics
- Motivational Interviewing (MI) (Experimental)
  Interventions: Behavioral: Motivational Interviewing
- Screening and Referral (S&R) (Active Comparator)
  Interventions: Behavioral: Screening and Referral

INTERVENTIONS:
Behavioral: Kisoboka — Intervention activities:
  Financial goal setting (developing delayed rewards), Text message reminders of savings goals (increase salience of delayed rewards), Substance-free activities (alternative reinforcers), Mobile money savings and work payments (constraints on buying alcohol), Social support & role models for financial goals and substance-free activities (delayed rewards, alternative reinforcers), Financial literacy, Develop motivation & confidence for change, Goal setting for alcohol reduction & ART adherence, Alcohol harms & defining low risk drinking Discuss challenges to change and maintain alcohol risk reduction and improved adherence, Developing & reinforcing discrepancy between savings/life goals and drinking/poor adherence, Developing discrepancy activity: goals for savings and healthy living and weekly, monthly, yearly spending on alcohol Self-monitoring of savings & spending Text message reminders to reinforce discrepancy between unhealthy behavior & goals
  Arms: Kisoboka (BE + MI and synergy)
Behavioral: Behavioral Economics — Intervention activities:
  Financial goal setting (developing delayed rewards), Text message reminders of savings goals (increase salience of delayed rewards), Substance free activities (alternative reinforcers), Mobile money savings and work payments (constraints on buying alcohol/ decrease reward value of alcohol), Social support & role models for financial goals and substance free activities (delayed rewards, alternative reinforcers), Financial literacy
  Arms: Behavioral Economics (BE)
Behavioral: Motivational Interviewing — Intervention activities:
  Develop motivation and confidence for change, Specific goal setting for alcohol reduction and ART adherence, Alcohol harms & defining low risk drinking, Discuss challenges to change and to maintain alcohol risk reduction and improved adherence/care engagement
  Arms: Motivational Interviewing (MI)
Behavioral: Screening and Referral — Brief feedback on their Alcohol Use Disorders Identification Test (AUDIT) score per the AUDIT brief intervention manual, a referral for alcohol counseling, and brief guidance on the importance of HIV care engagement and adherence following the Ugandan Ministry of Health protocol. A referral coupon with details of the clinic name and location will be provided to each participant and participants will be asked to submit the referral note to the "alcohol and/or HIV counselor".
  Arms: Screening and Referral (S&R)

SUMMARY:
The investigators developed the Kisoboka ("It is possible") Intervention to address limitations of existing evidence-based interventions to optimize treatment as prevention among men living with HIV who drink alcohol at hazardous levels in "risk environments" such as fishing communities through reductions in hazardous alcohol use, improved adherence to HIV medications and achieving undetectable HIV viral loads.

Social and structural determinants unique to fishing communities interact to create a risk environment where hazardous drinking impedes adherence to HIV medications among men living with HIV, including prevalent social norms of drinking, drinking as a way of experiencing "reward" and connecting with others (e.g. in the context of transactional sex), stressful work conditions, a "live for today" outlook, and a cash-based economy with no traditional savings infrastructure leading to ease of daily expenditure on drinking and sex work. These social and environmental conditions result in high levels of alcohol misuse and HIV risk, poor HIV outcomes, and exacerbation of HIV-associated wellness comorbidities such as poor mental and subjective physical health and food insecurity.

The goal of this study is to learn if the intervention called Kisoboka works to help men in fishing communities reduce hazardous alcohol use, be better able to take the participants HIV medication as prescribed, and have undetectable HIV viral loads. The investigators will compare the Kisoboka intervention to a brief alcohol screening, adherence counseling, and referrals, and to components of the Kisoboka intervention.

Participants will attend intervention counseling sessions according to the study arm to which the participants are randomly assigned. The number of sessions ranges from 1 to 6 over 1 to 16 weeks and are individual only or both individual and group sessions.

ELIGIBILITY:
Inclusion Criteria:

1. living with HIV;
2. residing in a fishing community (on most days/nights);
3. AUDIT-C positive (≥4) indicating potential hazardous drinking;
4. >6 months since initial antiretroviral treatment (ART) initiation;
5. not planning to move from the area within the next 6 months;
6. have their own mobile phone and can be reached via phone.
7. an indicator of potential suboptimal treatment as prevention (TasP) either:

(i) last HIV viral load test (within 6 months) was detectable (>20) or (ii) last viral load test between 6 and 13 months ago was detectable (>20) and reports missing ≥2 ART doses in the past 2 weeks or (iii) a lack of viral load test results for the prior 13 months in clinic records and reports missing ≥2 ART doses in the past 2 weeks;

Exclusion Criteria:

1. visibly intoxicated at enrollment (eligible to enroll when not intoxicated);
2. does not speak Luganda or English;
3. currently receiving a majority of work payments via mobile money/digital payments;
4. participated in the Kisoboka pilot RCT;
5. unable to read basic Luganda or English

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 716 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Change in Phosphatidylethanol (PEth) From Baseline | 6 and 12 month follow up
  alcohol biomarker which correlates well with the volume of alcohol consumed over the prior 2-4 weeks
Number of Participants with very Hazardous Alcohol Use at Baseline, 6, and 12 Month Follow up | 6 and 12 month follow up
  Combined biomarker self-report outcome. Number of participants with phosphatidylethanol values ≥400ng/mL OR AUDIT-C scores ≥9. AUDIT-C is the Alcohol Use Disorder Identification Test - Concise.
Number of Participants With Optimal Antiretroviral (ART) Adherence at Baseline, 6 and 12 Month Follow up | 6 and 12 month follow up
  ART levels tested using blood biomarkers with cut points indicating 6 or more doses per week
Number of Participants with Undetectable HIV Viral Loads at baseline, 6, and 12 month follow up | 6 and 12 month follow up
  HIV viral load laboratory test results showing undetectable viral load per the assay used (e.g., <20, <40 copies/ml)

SECONDARY OUTCOMES:
Change in depressive symptoms from baseline | 6 and 12 month follow up
  self-reported symptoms of depression using a shortened version of the "Center for Epidemiologic Studies Depression Scale" adapted for the population based on prior scale adaptation and validation. Minimum and maximum expected values are 0- 39 with higher scores indicating more depressive symptoms.
Number of participants with optimal self-reported Antiretroviral Adherence at Baseline, 6 and 12 months | 6 and 12 month follow up
  Self-reported adherence to antiretroviral treatment using the Instrument for Retrospective Adherence which includes an estimate of the number of doses missed over the previous 30-days and two subjective ratings of adherence
Change in subjective physical health from baseline | 6 and 12 month follow up
  Physical health summary score from the "HIV Medical Outcomes Survey" scale (MOS-HIV) including subscales of physical function, pain, role function, as well as energy/fatigue, overall health, and social function. Values for each subscale are transformed to 0 to 100 scale to permit comparisons with higher scores indicating better subjective physical health.
Number of participants who are food secure at baseline, 6 months, and 12 months | 6 and 12 month follow up
  Food insecurity is assessed using the "Household Food Insecurity Access" scale which assesses the degree of food insecurity/security in resource-limited settings. Scale scores are categorized into 4 categories ranging from Food Secure to Severely Food Insecure.

OTHER OUTCOMES:
Change in delayed reward discounting from baseline | 6 and 12 month follow up
  Delay discounting to assess the extent to which participants respond to immediate vs. delayed rewards using a context-adapted version of the "Monetary Choice Questionnaire" (MCQ). The most frequently reported index from the MCQ is the k value, which reflects the hyperbolic discounting function most consistent across a given participant's choices. Higher K scores are indicative of greater delayed reward discounting.
Change in endorsement of alternative reinforcers from baseline | 6 and 12 month follow up
  Measures the reinforcement from alcohol-free vs alcohol-involved activities incorporating availability using a context-adapted version of the Reinforcement-Survey Substance Use Version
Change from baseline in endorsement of the reward value of alcohol | 6 and 12 month follow up
  The hypothetical Alcohol Purchase Task self-report measure adapted to Ugandan prices used to generate indices of the reward value of alcohol.
Change from baseline in motivation to change behavior | 6 and 12 month follow up
  Items adapted from Information, Motivation, Behavioral Skills measures of motivation for antiretroviral adherence, and items adapted from the Theory of Planned Behavior (attitudes, subjective norms, perceived behavioral control, and intentions) measures for reducing hazardous alcohol consumption

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Kiene, PhD, MPH, Principal Investigator — San Diego State University; Joseph KB Matovu, PhD, MHS, Principal Investigator — Makerere University
Locations (1):
- Makerere University Walter Reed Program, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share raw questionnaire data. For all data, all identifiable information will be removed and maintained in a secure file for future contact purposes, but Global Unique Identifiers (GUIDs) or pseudoGUIDs will be assigned through the National Institute of Mental Health (NIMH) Data Archive. All other de-identified scientific data (questionnaire datasets, results from biological specimens testing, will be both preserved and shared through NIAAA Data Archive repository.
  Study protocol for the randomized controlled trial and survey questionnaires will be made available through NIAAA Data Archive repository. This documentation will be provided in portable document format (PDF).
  Scientific data will be processed and analyzed in standard statistical analysis software (e.g., SPSS, MPLUS, SAS, and R).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Baseline data, such as demographics and self-reported data, that require no additional analyses will be submitted to the NIAAA Data Archive repository within 4 months after enrollment. Baseline laboratory test data will be added as it becomes available. After the study is complete and unmasked, the study team will submit all remaining data (follow-up data). Data will be shared with the general research community at the time of an associated publication, or the end of the award/support period, whichever comes first. As required by NIAAA Data Archive repository, for each publication developed, the investigators will also create studies that contain the data used in that analysis and include the digital object identifiers (DOI) for that study (from NIAAA Data Archive repository) in the manuscript to aid in findability. NIAAA Data Archive repository makes determinations regarding how long to preserve the data; to date files have been preserved in perpetuity.
Access Criteria: Data will be findable for the research community through the NIMH Data Archive (NIAAA Data Archive specifically) which is established at the time of study funding. For all publications, an NIAAA Data Archive study will be created. Each of those studies is assigned a digital object identifier (DOI). This data DOI will be referenced in the publication. Investigators at institutions with a Federal Wide Assurance (FWA) will be able to gain access to NIAAA Data Archive repository data by submitting a data access request in accordance with applicable NIAAA Data Archive repository policies. Data requests will be reviewed and granted by an NIMH/NIAAA Data Archive Data Access Committee.
URL: https://nda.nih.gov/nda/access-data-info